CLINICAL TRIAL: NCT07093840
Title: Effectiveness of AmblyoPlay-Based Multimodal Therapy in Children With Anisometropic Amblyopia
Brief Title: Multimodal Therapy in Anisometropic Amblyopia
Acronym: MUTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yusa Basoglu (Other)
Collaborators: Smartoptometry (Unknown); Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor-Investigator, Yusa Basoglu, Istanbul Medipol University, Medipol University
Organization: Medipol University (Other)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-5860
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Amblyopia, Anisometropic; Pediatric; Postural Balance; Vision Therapy; Oculomotor System
Keywords: amblyopia; anisometropia; digital therapy; visual acuity; stereopsis; oculomotor function; motor skills; postural- balance
MeSH Terms: conditions — Amblyopia; Anisometropia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two parallel groups in a non-randomized manner: an intervention group that received AmblyoPlay-based visual therapy for 6 months, and a control group that did not receive any intervention. Group assignment was based on participant availability and preference. Both groups were assessed at baseline, 1st, 3 months, and 6 months using standardized visual, oculomotor, and balance measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: AmblyoPlay Digital Visual Therapy — AmblyoPlay is a home-based, app-delivered multimodal visual therapy program designed for children with amblyopia. The therapy consisted of 30-minute sessions, performed 5 days per week over a 6-month period. Exercises included gamified visual tasks targeting oculomotor control, visual acuity, stereopsis, visual-motor integration, and postural coordination. The software automatically adjusted task difficulty based on individual performance. Therapy was performed on a tablet or computer with red-green anaglyph glasses provided to participants
  Other Names: AmblyoPlay,; AmblyoPlay Vision Therapy; Multimodal Visual Therapy
Other: control group — Participants in this group were healthy children who did not receive any therapeutic intervention during the 6-month study period. They were age- and gender-matched with participants in the intervention group to ensure baseline comparability. Assessments were performed only at baseline and at the 6-month follow-up and included measurements of visual acuity, oculomotor function, stereopsis, visual-motor integration, and postural control.

SUMMARY:
This study aims to evaluate whether a six-month app-based visual therapy program, called AmblyoPlay, can improve visual acuity, oculomotor skills, and balance in children with anisometropic amblyopia (a type of "lazy eye" caused by unequal refractive errors between the eyes). The therapy uses interactive games to train visual and motor functions. The study compares children who receive this therapy with a control group of children who do not receive any intervention. Researchers aim to explore the effectiveness of a multidisciplinary, technology-assisted approach that addresses visual and sensorimotor functions through an integrated, child-centered perspective.

DETAILED DESCRIPTION:
This study investigates the effects of a six-month, app-based multimodal visual therapy program-AmblyoPlay-on visual acuity, oculomotor skills, hand-eye coordination, and postural control in children diagnosed with anisometropic amblyopia. Unlike traditional approaches that focus solely on monocular visual improvement, this study adopts a multidimensional, integrative framework that engages both visual and sensorimotor systems through gamified, child-friendly digital exercises.

The intervention is grounded in principles of dichoptic stimulation and neuroplasticity, aiming to reduce interocular suppression while promoting binocular cooperation. Through real-time adaptive difficulty algorithms, AmblyoPlay delivers personalized visual-motor challenges tailored to the developmental level of each participant.

Assessments are conducted at multiple time points to track progression across visual, motor, and postural domains. A control group of age- and sex-matched children with normal development is used for comparative analysis.

This study is designed to contribute evidence on the feasibility and efficacy of a multidisciplinary therapeutic model for pediatric amblyopia, highlighting the importance of addressing not only visual deficits but also associated functional impairments in balance and coordination.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 13 years

Diagnosed with anisometropic amblyopia according to AAO (American Academy of Ophthalmology) guidelines

No vestibular pathology within the past 6 months

No cognitive or mental impairments

No history of prior ophthalmologic treatment for amblyopia

Able to adhere to the treatment protocol

Written informed consent obtained from a parent or legal guardian

Exclusion Criteria:

* Age outside the range of 7 to 13 years

Presence of strabismus or other ocular pathologies (e.g., cataract, retinal disease)

Diagnosed neurological, developmental, or psychiatric disorders

Use of medications that may affect vision or balance

Participation in another clinical trial within the past 6 months

Inability to attend scheduled follow-up evaluations or comply with study procedures

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Baseline, 1 month, 3 months, and 6 months
  Visual acuity (VA) was assessed using a standard Snellen chart under both monocular and binocular viewing conditions. Participants were instructed to read optotypes from a distance of 6 meters for distance vision and 40 cm for near vision. Each eye was tested separately, followed by binocular testing. The smallest optotype correctly identified was recorded as the VA score. Results were documented in Snellen fractions and converted to decimal values for statistical analysis (e.g., 20/20 = 1.0; 20/40 = 0.5; 20/100 = 0.2). Higher decimal values represented better visual acuity.

SECONDARY OUTCOMES:
Stereopsis (Stereoacuity) | Baseline, 1 month, 3 months, and 6 months
  Stereoscopic vision was assessed using the Titmus Stereo Test. Participants wore polarized glasses and viewed the test booklet from a distance of approximately 40 cm. The test required identification of three-dimensional figures, including the fly, animal shapes, and Wirt circles. The stereoacuity threshold was recorded in arc seconds (arc-sec) based on the smallest disparity level correctly perceived. Scores were categorized as gross stereopsis (3600 arc-sec), moderate stereoacuity (800-200 arc-sec), and fine stereoacuity (100-40 arc-sec). Lower arc-sec values indicated better depth perception.

OTHER OUTCOMES:
Oculomotor Function | Baseline, 1 month, 3 months, and 6 months
  Oculomotor function was assessed through clinical observation of saccadic eye movements, smooth pursuit tracking, and fixation stability. Participants were asked to follow visual targets in various directions to evaluate the speed, accuracy, and coordination of eye movements. Abnormalities were noted using qualitative grading criteria. Assessments were conducted under standardized conditions at all time points.
Postural Stability (Sensory Organization Test - CDP) | Baseline, 1 month, 3 months, and 6 months
  Postural stability was assessed using the Sensory Organization Test (SOT) module of the computerized dynamic posturography (CDP) system. The test evaluated balance control under six sensory conditions by measuring sway and equilibrium scores. Participants stood barefoot on a force platform while visual and somatosensory inputs were altered. Composite and condition-specific balance scores were recorded. Higher scores indicated better postural stability.
Visual-Motor Integration (BOT-2) | Baseline, 1 month, 3 months, and 6 months
  Visual-motor integration skills were evaluated using selected subtests from the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2). Subtests included fine motor precision, fine motor integration, and manual coordination. Participants performed drawing, tracing, and object manipulation tasks. Standardized scores were calculated and compared across time points to assess changes in visual-motor performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, BEYKOZ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results reported in this study (after de-identification) will be made available to researchers upon reasonable request. Data will be shared for the purpose of academic research, including meta-analyses, and must be supported by a methodologically sound proposal. Access to the data will be granted beginning 6 months after publication and will remain available for 5 years. A data dictionary defining each variable will also be provided. Requests should be directed to: ybasoglu@medipol.edu.tr.
Supporting Information: SAP
Time Frame: IPD will be available beginning 6 months after publication of the primary manuscript and will remain available for 5 years.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to the de-identified individual participant data (IPD), including the study protocol, statistical analysis plan, informed consent form, and analytic code. Requests must be submitted via email to the principal investigator at ybasoglu@medipol.edu.tr. Each request will be reviewed for scientific merit and compliance with ethical standards. A data use agreement may be required prior to access.